CLINICAL TRIAL: NCT02802371
Title: Evaluation of the Impact of Personalized Pharmaceutical Collaborative Care Integrated to a Multidisciplinary Psychosocial Program on the Burden Felt by Caregivers of Elderly Patients With Alzheimer's Disease and Related Disorders and Evaluated at 18-month Follow-up
Brief Title: Pharmaceutical Collaborative Care Integrated to a Multidisciplinary Psychosocial Program
Acronym: PHARMAID
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 69HCL14_0450
Record Dates: First submitted 2016-06-08; First posted 2016-06-16 (Estimated); Last update posted 2019-01-10 (Actual); Status verified 2019-01

CONDITIONS: Alzheimer Disease
Keywords: caregiver burden; Alzheimer disease and related disorders; elderly; pharmaceutical care; optimization of drug prescribing; psychosocial intervention
MeSH Terms: conditions — Alzheimer Disease; Caregiver Burden | interventions — Psychosocial Intervention; Pharmaceutical Services; Psychiatric Rehabilitation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- control group (No Intervention): Patients and caregivers randomized in the control group will receive the current management in geriatric or memory consultation without multidisciplinary psychosocial intervention and pharmaceutical collaborative care.There will be a history of the drugs prescribing leading to pharmaceutical recommendations by the pharmacist-clinician, but the recommendations will not be transmitted to the referring physicians of patients and caregivers.
- Psychosocial intervention (Active Comparator): Psychosocial intervention including collective sessions and individual interview in face-to-face and by phone. These sessions will allow an extended psychosocial follow-up over one year.
  Interventions: Behavioral: Psychosocial intervention
- Pharmaceutical care and psychosocial support (Experimental): Pharmaceutical collaborative care integrated in a psychosocial program. The clinical pharmacist will intervene in: 1) the pharmaceutical need assessment of caregivers; 2) collective session on medication management; and 3) optimization of drug prescribing. These collective and individual sessions of pharmaceutical care will allow an extended 18 month follow-up. Psychosocial intervention including collective sessions and individual interview in face-to-face and by phone. These sessions will allow an extended psychosocial follow-up over one year.
  Interventions: Other: Pharmaceutical care and psychosocial support

INTERVENTIONS:
Behavioral: Psychosocial intervention — Caregivers included in this group will benefit from a multi-component intervention with three collective sessions and individual interview in face-to-face or by phone according to the follow-up time.
  Arms: Psychosocial intervention
Other: Pharmaceutical care and psychosocial support — Caregivers included in this group will benefit from the same multi-component intervention that group "psychosocial intervention" with the integration of pharmaceutical care by a clinical pharmacist. The clinical pharmacist will intervene in: 1) the pharmaceutical need assessment of the caregivers considering their medication management and the medication management of their relatives at the inclusion; 2) a collective session on medication management; and 3) personalized interviews to consider needs, medication problems and difficulties in the therapeutic optimization process.
  Arms: Pharmaceutical care and psychosocial support

SUMMARY:
Caring for patients with Alzheimer Disease or Related Disorders (ADRD) is accompanied with a caregiver burden that increases with the progression of the disease. This burden can have physical, psychological, emotional, social and financial issue on the informal caregivers who are often represented as hidden secondary patients. They frequently have a higher risk of developing mood disorders as depression, anxiety, stress, sleep disorders and a lower quality of life associated with a greater use of psychotropic drugs. They also incur higher risk of heart disease and mortality. The embrittlement of the caregiver is a major factor of early institutionalization of patient. In the PIXEL study, the mean age of the men caregivers was 73.9 years and 64.8 for the women caregivers. Elderly themselves, especially spouses, the informal caregivers are also exposed to common chronic diseases and associated polypharmacy with a higher risk of developing drug-related problems due to aging and negligence of their own health care. These risks are increased mainly in the elderly because of changes in pharmacokinetic and pharmacodynamic parameters related to aging, acute or chronic diseases and the potentially inappropriate prescription (PIP). Previous studies have shown the effectiveness and positive impact of optimization of the therapeutics by a clinical pharmacist on the reduction of drug-related problems, length of hospital stay, readmission rates, quality of life and mortality. The patient's medication management is usually delegated to the informal caregiver, who must also manage his own treatment. The caregiver may face difficulties with therapeutics (e.g., inappropriate dosage form, adverse effects and patient refusal) that could impact on its compliance with treatment or that of his relative. No previous study has evaluated the impact of pharmaceutical collaborative care including personalized interview with a clinical pharmacist and optimization of drug prescribing among patients with ADRD and their caregivers.

However, many studies have assessed the effectiveness of non-pharmacological interventions on caregiver burden, mood disorders and the patient institutionalization. Meta-analysis showed a moderate improvement of the caregiver burden.

The main objective of the PHARMAID study is to measure the impact of personalized pharmaceutical collaborative care integrated to a multidisciplinary psychosocial program on the burden of ADRD caregivers and assessed at 18-month follow-up.

ELIGIBILITY:
Inclusion Criteria:

for the patients:

* Patients aged 65 and over;
* Patients with ADRD;
* Patients suffering from mild to moderate stages of the disease, defined by the Mini-Mental Score Examination (MMSE), with scores of 25 to 16/30;
* Patients living at home;
* Patients received in a geriatric or memory consultation of a study recruiting centers;
* Patients with the ability to express themselves orally or in writing in French sufficiently to carry out clinical assessments;
* Patients who are not opposed to the research;

for the caregivers:

* Caregivers aged 55 and over;
* Nonprofessional caregivers living with the patient or providing support to him/her at least 10 hours a week for the activities of daily living;
* Caregivers with the ability to follow the program at the discretion of the investigator;
* Caregivers with the ability to express themselves orally or in writing in French sufficiently to carry out clinical assessments;
* Caregivers who are not opposed to the research.

Exclusion Criteria:

for the patients:

* Institutionalized patients.

for the caregivers:

* Caregivers involved in another support program for the caregivers;
* Caregivers whose the level of acceptance of the disease does not allow the participation in the study.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2016-08 (Actual); Primary Completion 2020-02 (Estimated); Study Completion 2020-02 (Estimated)

PRIMARY OUTCOMES:
caregiver's burden | Change from Baseline at 18-months follow-up
  The caregiver burden is measured using the Zarit Burden Index (ZBI) questionnaire. The ZBI is a subjective measure of burden that includes 22 items exploring the caregiver's perception and feelings about care situations. Each item was evaluated using a 5-point Likert scale ranging from 0 (never) to 4 (almost always), which are summed. The score range is 0-88, a higher score indicating a higher burden level.

SECONDARY OUTCOMES:
caregiver's quality of life | Change from Baseline at 18-months follow-up
  Quality of life measured by questionnaire EUROQOL 5D
caregiver's anxiety | Change from Baseline at 18-months follow-up
  anxiety measured by scale HARD
caregiver's depression | Change from Baseline at 18-months follow-up
  depression measured by Geriatric Depression Scale (GDS)
patient's quality of life | Change from Baseline at 18-months follow-up
  Quality of life measured by questionnaire Alzheimer Disease Related Quality of Life (ADRQL scale)
patient's behavioral disorders | Change from Baseline at 18-months follow-up
  behavioral disorders measured by questionnaire Neuropsychiatric Index (NPI)
patient's functional autonomy | Change from Baseline at 18-months follow-up
  functional autonomy measured by IADL scale (Instrumental Activities of Daily Living)
Occurrence of medical consultation | Change from Baseline at 18-months follow-up
  number of medical consultation in patients and caregivers
Occurrence of recourse to emergency service | Change from Baseline at 18-months follow-up
  occurrence of recourse to emergency service in patients and caregivers
Occurrence of hospitalizations | Change from Baseline at 18-months follow-up
  number of hospitalization in patients and caregivers
Occurrence of admission in institution | Change from Baseline at 18-months follow-up
  occurrence of admission in institution in patients

CONTACTS AND LOCATIONS:
Overall Officials: Christelle Mouchoux, PharmD, PhD, Principal Investigator — Pharmacy unit and Clinical Research Center VCF (" Aging Brain Frailty ") University hospital of Lyon, Charpennes Hospital / University Lyon / INSERM, U1028; CNRS, UMR5292; Lyon Neuroscience Research Center, Lyon, France.
Locations (1):
- Pharmacy unit and Clinical Research Center VCF (" Aging Brain Frailty ") University hospital of Lyon, Charpennes Hospital / University Lyon / INSERM, U1028; CNRS, UMR5292; Lyon Neuroscience Research Center, Villeurbanne, France

REFERENCES:
- [Derived] Novais T, Qassemi S, Cestac P, McCambridge C, Villars H, Zueras A, Decaudin B, Dambrine M, Huvent-Grelle D, Roche J, Schoenenburg S, Federico D, Nier AC, Krolak-Salmon P, Mouchoux C. Impact of pharmaceutical care integrated at a psychosocial intervention to reduce caregiver's burden in Alzheimer's disease or related dementias: Negative results at 18 months and difficulties to conduct PHARMAID RCT. Contemp Clin Trials Commun. 2023 Apr 22;33:101146. doi: 10.1016/j.conctc.2023.101146. eCollection 2023 Jun. PMID 37397433
- [Derived] Novais T, Moutet C, Delphin-Combe F, Dauphinot V, Colin C, Krolak-Salmon P, Mouchoux C; PHARMAID study group. PHARMAID study protocol: Randomized controlled trial to assess the impact of integrated pharmaceutical care at a psychosocial intervention on caregiver's burden in Alzheimer's disease or related diseases. Contemp Clin Trials. 2017 Feb;53:137-142. doi: 10.1016/j.cct.2016.12.020. Epub 2016 Dec 19. PMID 28007635